CLINICAL TRIAL: NCT05775185
Title: Changes in Therapeutic Response, Ocular Manifestations of Graves' Orbitopathy and Quality of Life During the First Year After Orbital Radiotherapy
Brief Title: Therapeutic Efficacy of Orbital Radiotherapy in Patients With Graves' Orbitopathy
Status: Completed | Type: Observational
Sponsor: Medical University of Sofia (Other)
Responsible Party: Principal Investigator, Mariya Stoynova, Principal investigator, Medical University of Sofia
Other Study IDs: 21B /25.07.2017
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Orbital radiotherapy: The study includes only one group of patients treated with orbital radiotherapy for 2-week period, a total dose of 20 Gy, 2Gy for each session.
  Interventions: Radiation: Orbital radiotherapy

INTERVENTIONS:
Radiation: Orbital radiotherapy — Low dose fractionated orbital radiotherapy, total dose 20 Gy in 2-week period.

SUMMARY:
The purpose of the present interventional study is to assess the changes in the therapeutic response, ocular manifestations of Graves' orbitopathy and quality of life during the first year after orbital radiotherapy. The main questions it aim to answer are:

1. How effective is orbital radiotherapy used as first- or second-line treatment in patients with Graves' orbitopathy?
2. How does the quality of life changes after orbital radiotherapy?

Participants have active moderate-to-severe Graves' orbitopathy and are treated with low dose fractionated orbital radiotherapy for two weeks. During the follow-up period they undergo regular ocular examinations and fill out a disease-specific questionnaire.

DETAILED DESCRIPTION:
Orbital radiotherapy is a well-established second-line therapy for moderate-to-severe forms of Graves' orbitopathy. However, the question about it efficacy is still controversial. The purpose of the present interventional study is to assess the changes in the therapeutic response, ocular manifestations of Graves' orbitopathy and quality of life during the first year after orbital radiotherapy. The main questions it aim to answer are:

1. How effective is orbital radiotherapy used as first- or second-line treatment in patients with Graves' orbitopathy?
2. How does the quality of life changes after orbital radiotherapy?

Participants have active moderate-to-severe Graves' orbitopathy untreated or already treated with systemic glucocorticoids and are referred to low dose fractionated orbital radiotherapy, total dose 20 Gy divided into 10 sessions, 2 Gy for each session. A concomitant intake of low-dose glucocorticoids is prescribed to all patient. During the follow-up period they undergo regular ocular examinations (at 1st, 3rd, 6th and 12th month), which includes comprehensive ocular status, hormonal and immunological testing and evaluation of the current therapeutic response. The patients also fill out a disease-specific questionnaire (at 3rd, 6th and 12th months).

ELIGIBILITY:
Inclusion Criteria:

- Active moderate-to-severe Graves' orbitopathy

Exclusion Criteria:

* Contraindications for orbital radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 26 patients with active moderate-to-severe Graves' orbitopathy. Eight of them have untreated disease and the rest have been already treated with systemic glucocorticoids. Patients with contraindications for orbital radiotherapy are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Efficacy of orbital radiotherapy | 12 months
  Effect on therapeutic response and individual ocular parameters
Effect of orbital radiotherapy on quality of life | 12 months
  Effect of orbital radiotherapy on disease-specific quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mariya A Stoynova, Principal Investigator — Medical University of Sofia: Medicinski universitet-Sofia
Locations (1):
- University Hospital of Endocrinology, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stoynova MA, Shinkov AD, Novoselski MT, Petrova VV, Dimitrova ID, Yankova IA, Kovatcheva RD. Changes in therapeutic response, ocular manifestations of Graves' orbitopathy and quality of life during the first year after orbital radiotherapy. Int Ophthalmol. 2023 Nov;43(11):4305-4314. doi: 10.1007/s10792-023-02842-8. Epub 2023 Aug 10. PMID 37561249